CLINICAL TRIAL: NCT02599064
Title: A Phase 1/2 Multicenter, Multidose, Dose Escalation Study to Evaluate the Safety, Tolerability and Clinical Activity of RXI-109 Administered by Intravitreal Injection to Reduce the Progression of Subretinal Fibrosis in Subjects With Advanced Neovascular Age-related Macular Degeneration
Brief Title: Evaluating RXI-109 to Reduce the Progression of Subretinal Fibrosis in Subjects With NVAMD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RXi Pharmaceuticals, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXI-109-1501
Record Dates: First submitted 2015-11-03; First posted 2015-11-06 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Age-related Macular Degeneration; Subfoveal Choroidal Neovascularization; Subretinal Scarring; Subretinal Fibrosis
Keywords: Age-related macular degeneration; RXI-109; NVAMD; Retinal scarring; Subretinal scarring; Retinal fibrosis; Subretinal fibrosis; Eye diseases
MeSH Terms: conditions — Macular Degeneration; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RXI-109 (Experimental): Intravitreal injections of RXI-109 in one eye given on Day 1 and at monthly intervals through Month 3 for a total of four doses
  Interventions: Drug: RXI-109

INTERVENTIONS:
Drug: RXI-109 — RXI-109 dosed intravitreally to subjects with NVAMD

SUMMARY:
This study is designed to evaluate the safety, tolerability and clinical activity of RXI-109 administered by intravitreal injection to reduce the progression of subretinal fibrosis in subjects with advanced neovascular age-related macular degeneration (NVAMD).

DETAILED DESCRIPTION:
Evaluate the safety, tolerability and pharmacokinetics (PK) of single and multiple doses of RXI-109 when administered by intravitreal injection. Evaluate the clinical activity of single and multiple doses of RXI-109 when administered by intravitreal injection. Study participation is intended to be seven months from time of initial treatment with RXI-109.

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting with advanced NVAMD in the study eye with BCVA ≤20/100 potentially due to subretinal fibrosis involving the fovea
* BCVA ≥20/800 in the contralateral eye and better than the study eye
* ≥50 years of age
* Subfoveal choroidal neovascularization (CNV) of any type

Exclusion Criteria:

* Presence of other causes of CNV including pathologic myopia, ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, and multifocal choroiditis
* Evidence of inflammation (Grade 1 or higher) in the anterior or posterior chamber

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and relationship of AEs, including clinically significant changes in physical examination findings, ocular examinations and assessments, and clinical laboratory results | Seven (7) months
  Assess severity and frequency of reported adverse events graded by CTCAE, ophthalmological exams to assess clinically relevant changes in ocular health, clinically-relevant changes in physical exams or laboratory testing assessed by medical personnel, and monitoring for any change in best corrected visual acuity (BCVA)
Pharmacokinetic profile of RXI-109 in blood | Four (4) months
  Determine systemic exposure (AUC) of RXI-109 after intra-ocular injections

SECONDARY OUTCOMES:
Relative change (%) of subretinal fibrosis lesion size compared to baseline using standard ophthalmologic imaging. | Seven (7) months
  Evaluate the clinical activity of RXI-109 to reduce the formation or progression of subretinal fibrosis
Changes from baseline in BCVA using the Early Treatment Diabetic Retinopathy (ETDRS) chart | Seven (7) months
  Evaluate the clinical activity of RXI-109 by assessing changes in visual acuity

OTHER OUTCOMES:
Relative change (%) of CTGF protein levels in aqueous fluid compared to baseline | Seven (7) months
  Evaluate the clinical activity of RXI-109 by assessing changes in CTGF protein levels in aqueous fluid

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit Dispersyn, Study Director — RXi Pharmaceuticals
Locations (1):
- Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland, United States